CLINICAL TRIAL: NCT05593289
Title: Effectiveness of the Neck-Specific Exercise Program Through TeleRehabilitation Compared to the Usual Intervention in Functional Recovery in Adults With Acute Cervical Sprain Grade I and II in the First Level of Care
Brief Title: Effectiveness of a Telerehabilitation Program in Acute Cervical Sprain Grade I and II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Juan Figueroa-García, Principal investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2022-3511-021
Record Dates: First submitted 2022-10-18; First posted 2022-10-25 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Neck Sprain; Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): Participants assigned to the telerehabilitation program will complete a 3 month intervention consisting of 5 weekly sessions of 30 minutes of pre-recorded video, with a frequency of 2-3 times a day.
  Interventions: Other: telerehabilitation
- Control group (No Intervention): The usual care group will be instructed to follow their physicians' orders during the 3-month intervention period. Baseline measurements will be made for each group, at 2 weeks, 6 weeks and 3rd month.

INTERVENTIONS:
Other: telerehabilitation — Physical activity that is planned, structured with repeated muscle movements with the aim of relearning motor skills, resistance of neck muscles and postural correction.
  Arms: Telerehabilitation group

SUMMARY:
Cervical sprain also known as whiplash-associated disorder is the result of a combined injury between extension/flexion of the soft tissues of the cervical spine due to an acceleration-deceleration mechanism of energy transfer to the neck. The Neck-Specific Exercise Program focuses on relearning motor skills, neck muscle endurance, and postural correction. Telehealth improves patient satisfaction, overcomes barriers to access to physiotherapy services and reduces the costs of musculoskeletal care.

Objective: To evaluate the effectiveness of the neck specific exercise program by telerehabilitation compared to the usual intervention in functional recovery in adults with acute cervical sprain grade I and II at the first level of care.

Material and Methods: This is a randomized clinical trial, the effectiveness of the telerehabilitation program is determined by the Neck Disability Index (NDI) and will be compared against the usual intervention. Participants assigned to the telerehabilitation program will complete a 12-week intervention consisting of 5 weekly sessions of 30 minutes of pre-recorded video, with a frequency of 2-3 times a day. The usual care group will be instructed to follow their doctors' orders during the 12-week intervention period. For each group, baseline measurements were made at 2, 6 and 12 weeks.

Time to develop: The protocol has a duration of follow-up of the patients of 12 weeks.

DETAILED DESCRIPTION:
The neck-related musculoskeletal disorders (MSDs), whether attributed to work, injury, or other activities manifest neck pain, are a prevalent source of disability and a common reason for consulting primary health care providers, including physical therapists and primary care physicians. Neck pain related to disorders associated with cervical sprain is the most common result of car accidents. Associated cervical sprain disorders disrupt the daily lives of adults worldwide and are associated with considerable pain, suffering, disability and costs. Cervical sprain (CD), also known as whiplash-associated disorder, is the result of a combined extension/flexion injury of the soft tissues of the cervical spine due to an acceleration-deceleration mechanism of energy transfer to the neck. The Quebec Task Force Classification System, is the classification that determine the degree of injury. This classification is based solely on clinical signs, dividing them into 5 categories: 0. Asymptomatic, 1. Cervical pain, muscle spasm, no physical signs, 2. Stiffness, localized pain, 3. Symptoms, signs and neurological clinic and 4. Bone injury, fracture/dislocation.

The objective of treatment should be aimed at restoring the functionality of the individual with a biopsychosocial approach, so that structured patient education should be considered, making patients aware of the typical course and treatment of grade I-II CD, the importance of maintaining life activities and movement, to actively participate in your care plan by remaining active and maintaining neck movement, emphasizing active treatments instead of passive treatments. The main objective is to reincorporate the patient into daily life activities. Functionality is defined as: "the ability of the person to autonomously perform the activities of daily living." The loss of functionality in CD is associated with chronic pain, limitation in the arcs of movement, it is also an indicator of mental health. The effects of telerehabilitation, when associated with usual care or as an independent intervention, have also been evaluated in chronic non-malignant musculoskeletal pain. The use of telerehabilitation as a tool for conducting MSD assessments has been investigated, specifically in adults with non-specific neck pain compared to conventional methods, finding validity and reliability, thus adding more evidence to the existing evaluation based on telerehabilitation for MSDs.

Problem statement: In Mexico, the Mexican Institute of Social Security provides care for this type of condition, however in the Family Medicine Units (primary health) there are no physiotherapists who evaluate and manage the cervical sprain early which has been demonstrated, has an impact on the functional recovery time of patients with muscle injuries, the above is important since it has been shown that early rehabilitation is one of the most effective strategies for functional recovery in musculoskeletal disorders.

Research question: What is the effectiveness of the Neck-Specific Exercise Program by telerehabilitation compared to the usual intervention in functional recovery in adults with grade I and II acute cervical sprain at the first level of care?

Hypothesis: The effectiveness of the Neck-Specific Exercise Program in functional recovery in adults with grade I and II acute cervical sprain who performed the neck-specific exercise program using telerehabilitation for 6 weeks is that they will improve at least 3.5 points or more in levels of functionality through the Neck Disability Index (NDI) compared to those who performed the usual intervention.

Objective: To assess the effectiveness of the Neck-Specific Exercise Program though telerehabilitation compared with the usual intervention in functional recovery in adults with grade I and II acute cervical sprain at the first level of care.

Material and Methods Studio Design: This is a randomized clinical trial, in which the effectiveness of the telerehabilitation program is determined by the functionality indicator using the Neck Disability Index and will be compared against the usual intervention. Randomization will be carried out through the generation of random numbers in the Office Excel program by blocks of 5, to assignment to the experimental treatment and control will be carried out through opaque envelopes according to the distribution generated by computer, at the time of assignment to the treatment the researcher will not have any bias in assigning one or another treatment. The recruitment of participants, the assignment of participants to interventions and evaluations will be carried out by independent evaluators. Blinding of participants and staff in charge of teaching the telerehabilitation program as well as the usual intervention will not be possible due to the nature of the intervention. Evaluators will be blinded to group assignment as it will be other evaluators who assign participants to groups and conduct follow-up evaluations. Participants assigned to the telerehabilitation program will complete a 3-month intervention consisting of 5 weekly sessions of 30 minutes of pre-recorded video, with a frequency of 2-3 times a day. The usual care group will be instructed to follow your doctors' orders during the 3-month intervention period. For each group, baseline measurements will be made, at 2 weeks, 6 weeks and 12 weeks.

Sample Size: For the calculation of the sample size, it was based on the formula of the sample of an average. Considered a statistically significant difference in the Neck Disability Index to measure neck functionality, having a result of 3.5 (standard deviation 6.3), with a significance level of 0.05 and a power of 80%, an estimated loss of 20% is considered, a sample size of 28 subjects is estimated, plus the estimated loss a final sample of 34 subjects. Explicative variables: Specific Neck Exercise Program (NSE) through planned telerehabilitation physical activity. Outcome variables: Functional capacity of the neck, it will be obtained through the Neck Disability Index (NDI) and pain, it will be obtained through the Visual Analogue Scale.

Recruitment and Data Collection Process: Patients who present a first-time diagnosis of grade I and II cervical sprain will be selected from the consultation of the Family Medicine Unit number 33. Potential participants will be identified through a 5-step process, this process includes: 1. The study will be invited by direct invitation by the attending physician as well as posters placed in the offices and advertising areas within the clinic, once there is interest on the part of the patients, in a space specifically designated for the approach of the participants. 2. It will be make a check of medical records in case there is uncertainty or any missing data regarding the medical history. 3. Participants will be selected to determine their eligibility using the selection criteria. 4. It will perform a clinical physical examination performed by an experienced physician or physical therapist to classify the disorder as a grade I or II. 5.The participants will be given the NDI questionnaire for self-assessment.

Intervention neck-specific exercise program: All participants will receive verbal and written information about the study, once they accept and sign the informed concentration, they will be taught the use of the telerehabilitation program (which consists of written, graphic and video information on the digital platform, which is a teaching system designed to create and manage adapted online learning spaces) that they must make, as well as written information of the program, once they finish the teaching activity of the platform, emphasis will be placed on doubts about the use of the platform, in case of having any doubt, it will be resolved at that time. The telerehabilitation program is designed on a weekly basis, which will be explained to the participant the way in which they must do it. Once the teaching activity of use of the platform is finished, a resistance link will be given to the patient to be able to carry out a part of the protocol and will be followed up through it, since, through digital platform, you can know the time spent interacting with it; the time of the telerehabilitation activities will be 30 minutes daily.

The telerehabilitation program of Neck-Specific Exercise (NSE) is divided into 3 stages with a final duration of 12 weeks. The first stage consists of a series of three exercises, which will be performed isometric contractions maintained of five seconds with a rest between them of five seconds, which will be distributed in three series of five repetitions. It aims to facilitate deep muscle activity of the neck, without superficial muscle activity. The second stage consists of a series of three exercises, which will be performed resisted isometric contractions of five seconds of contraction with a rest between them of five seconds, which will be distributed in three series of 10 repetitions. The third stage consists of a series of five exercises, which will perform concentric contractions of progressive resistance, which will be distributed in three series of 20 repetitions. An initial face-to-face evaluation will be carried out (at study entry) and follow-up will be given for 12 weeks (by telephone at weeks 2, 6 and 12 after entering the study). Usual intervention: In the usual intervention the patient will be provided with the usual exercise program which contains a series of exercises that are routinely used to address this pathology, which must be performed three times a day, 10 times each, as well as an explanation of them and will be sent home for completion.

Descriptive statistics: The qualitative variables will be summarized in absolute and relative frequencies and the quantitative variables in measures of central tendency and dispersion, if they meet the criterion of normality by means of the Kolmogorov-Smirnov test will be used mean and standard deviation in case of not fulfilling the assumption will be used median and quartile 1 and 3. Inferential statistics: For the comparison of the dependent variables in the telerehabilitation group, before and at the end of the study student's t will be used for related samples , if they do not meet the normality criterion, the Wilcoxon test will be used. In order to identify possible confounding variables, the clinical and demographic characteristics will be compared, to compare the quantitative variables, student's t will be used and McNemar's Chi square will be used to compare the qualitative variables. A value of p< 0.05 shall be considered statistically significant. All analyses will be performed using the statistical program Stata version 14.

Ethical Considerations: The present protocol that will be carried out in the adult population with acute cervical sprain grade I and II, this adheres to the guidelines of the Declaration of Helsinki and those of the Mexican General law of health in force about research in human beings. Confidentiality: The data provided in this study are totally confidential, their results will be used globally and for statistical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients of the Mexican Social Security Institute of both sexes between 18-60 years old.
* That they are diagnosed with grade I or II acute cervical sprain for the first time Agree to participate in the study and sign the informed consent.
* That they are users of smartphone and / or computer with internet connection.
* Have the approval of the attending physician.

Exclusion Criteria:

* Not knowing how to read or write.
* Patients with neurological conditions.
* Loss of alertness or memory during the event that generated the cervical sprain.
* History of cervical disc herniations, nerve compressions with cervical irradiation, myelopathy, cervical surgeries, fibromyalgia.
* Allergy to latex.
* Patients whose work activity is considered by the attending physician as very heavy.

Elimination Criteria:

* Failure to complete the evaluation instrument in its entirety
* Failure to complete the telerehabilitation program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-11-17 (Estimated); Study Completion 2023-11-24 (Estimated)

PRIMARY OUTCOMES:
Changes in neck functionality, from baseline and at weeks 2, 6 and 12 | A baseline measurement at study entry, then three more follow-up assessments at week 2, week 6, and 12 weeks
  Ability of the person in his neck to perform activities of daily living, which will be measured with the Neck Disability Index (NDI), which scores from 0 to 50 points, where 0 is poor neck functionality and 50 is better functionality.

SECONDARY OUTCOMES:
Changes in neck pain, from baseline and at weeks 2, 6 and 12 | A baseline measurement at study entry, then three more follow-up assessments at week 2, week 6, and 12 weeks
  An unpleasant sensation induced by noxious stimuli which are detected by nerve endings of nociceptive neurons, which will be measured with the analog scale of pain, which has a score of 0 to 10, where 0 is no pain and 10 is the maximum pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Juan Figueroa, MSc, Principal Investigator — Juan Figueroa
Locations (2):
- Mexico (2):
  - Unidad de Medicina Familiar 21, Iztacalco, Mexico City
  - Unidad de Medicina Familiar 21, Mexico City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark P, Denova-Gutierrez E, Razo C, Rios-Blancas MJ, Lozano R. The burden of musculoskeletal disorders in Mexico at national and state level, 1990-2016: estimates from the global burden of disease study 2016. Osteoporos Int. 2018 Dec;29(12):2745-2760. doi: 10.1007/s00198-018-4698-z. Epub 2018 Sep 21. PMID 30242448
- [Background] Yelin E, Weinstein S, King T. An update on the burden of musculoskeletal diseases in the U.S. Semin Arthritis Rheum. 2019 Aug;49(1):1-2. doi: 10.1016/j.semarthrit.2019.04.010. Epub 2019 May 2. No abstract available. PMID 31133279
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Bussieres AE, Stewart G, Al-Zoubi F, Decina P, Descarreaux M, Hayden J, Hendrickson B, Hincapie C, Page I, Passmore S, Srbely J, Stupar M, Weisberg J, Ornelas J. The Treatment of Neck Pain-Associated Disorders and Whiplash-Associated Disorders: A Clinical Practice Guideline. J Manipulative Physiol Ther. 2016 Oct;39(8):523-564.e27. doi: 10.1016/j.jmpt.2016.08.007. PMID 27836071
- [Background] Spitzer WO, Skovron ML, Salmi LR, Cassidy JD, Duranceau J, Suissa S, Zeiss E. Scientific monograph of the Quebec Task Force on Whiplash-Associated Disorders: redefining "whiplash" and its management. Spine (Phila Pa 1976). 1995 Apr 15;20(8 Suppl):1S-73S. No abstract available. PMID 7604354
- [Background] Luan F, Yang KH, Deng B, Begeman PC, Tashman S, King AI. Qualitative analysis of neck kinematics during low-speed rear-end impact. Clin Biomech (Bristol). 2000 Nov;15(9):649-57. doi: 10.1016/s0268-0033(00)00031-0. PMID 10946097
- [Background] Sterling M. Physiotherapy management of whiplash-associated disorders (WAD). J Physiother. 2014 Mar;60(1):5-12. doi: 10.1016/j.jphys.2013.12.004. Epub 2014 Apr 24. No abstract available. PMID 24856935
- [Background] Bunketorp L, Lindh M, Carlsson J, Stener-Victorin E. The effectiveness of a supervised physical training model tailored to the individual needs of patients with whiplash-associated disorders--a randomized controlled trial. Clin Rehabil. 2006 Mar;20(3):201-17. doi: 10.1191/0269215506cr934oa. PMID 16634339
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Mani S, Sharma S, Singh DK. Concurrent validity and reliability of telerehabilitation-based physiotherapy assessment of cervical spine in adults with non-specific neck pain. J Telemed Telecare. 2021 Feb;27(2):88-97. doi: 10.1177/1357633X19861802. Epub 2019 Jul 4. PMID 31272309
- [Background] Wiangkham T, Duda J, Haque MS, Price J, Rushton A. A cluster randomised, double-blind pilot and feasibility trial of an active behavioural physiotherapy intervention for acute whiplash-associated disorder (WAD)II. PLoS One. 2019 May 9;14(5):e0215803. doi: 10.1371/journal.pone.0215803. eCollection 2019. PMID 31071100
- [Background] Bring A, Asenlof P, Soderlund A. What is the comparative effectiveness of current standard treatment, against an individually tailored behavioural programme delivered either on the Internet or face-to-face for people with acute whiplash associated disorder? A randomized controlled trial. Clin Rehabil. 2016 May;30(5):441-53. doi: 10.1177/0269215515581503. Epub 2015 Apr 20. PMID 25896985
- [Background] Gialanella B, Ettori T, Faustini S, Baratti D, Bernocchi P, Comini L, Scalvini S. Home-Based Telemedicine in Patients with Chronic Neck Pain. Am J Phys Med Rehabil. 2017 May;96(5):327-332. doi: 10.1097/PHM.0000000000000610. PMID 27584139
- [Background] Peolsson A, Landen Ludvigsson M, Overmeer T, Dedering A, Bernfort L, Johansson G, Kammerlind AS, Peterson G. Effects of neck-specific exercise with or without a behavioural approach in addition to prescribed physical activity for individuals with chronic whiplash-associated disorders: a prospective randomised study. BMC Musculoskelet Disord. 2013 Oct 30;14:311. doi: 10.1186/1471-2474-14-311. PMID 24171699
- [Background] Maramba I, Chatterjee A, Newman C. Methods of usability testing in the development of eHealth applications: A scoping review. Int J Med Inform. 2019 Jun;126:95-104. doi: 10.1016/j.ijmedinf.2019.03.018. Epub 2019 Mar 31. PMID 31029270
- [Background] Harte R, Glynn L, Rodriguez-Molinero A, Baker PM, Scharf T, Quinlan LR, OLaighin G. A Human-Centered Design Methodology to Enhance the Usability, Human Factors, and User Experience of Connected Health Systems: A Three-Phase Methodology. JMIR Hum Factors. 2017 Mar 16;4(1):e8. doi: 10.2196/humanfactors.5443. PMID 28302594
- [Background] Rothgangel A, Braun S, Smeets R, Beurskens A. Design and Development of a Telerehabilitation Platform for Patients With Phantom Limb Pain: A User-Centered Approach. JMIR Rehabil Assist Technol. 2017 Feb 15;4(1):e2. doi: 10.2196/rehab.6761. PMID 28582249
- [Background] Walton DM, Elliott JM. An Integrated Model of Chronic Whiplash-Associated Disorder. J Orthop Sports Phys Ther. 2017 Jul;47(7):462-471. doi: 10.2519/jospt.2017.7455. Epub 2017 Jun 16. PMID 28622487
- [Background] Hernandez-Sousa MG, Sanchez-Avendano ME, Solis-Rodriguez A, Yanez-Estrada M. [Disability by cervical sprain I and II and the use of neck collar]. Rev Med Inst Mex Seguro Soc. 2013 Mar-Apr;51(2):182-7. Spanish. PMID 23693107
- [Background] Chen HB, Yang KH, Wang ZG. Biomechanics of whiplash injury. Chin J Traumatol. 2009 Oct;12(5):305-14. PMID 19788851